CLINICAL TRIAL: NCT04585685
Title: Healthy Recovery After Trauma Study
Acronym: HRT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Christal L Badour (Other)
Responsible Party: Sponsor-Investigator, Christal L Badour, Assistant Professor of Psychology, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 59226
Record Dates: First submitted 2020-10-06; First posted 2020-10-14 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Stress Disorders, Post-Traumatic; Shame; Guilt; Sexual Assault and Rape
Keywords: post-traumatic stress disorder; mental contamination; cognitive processing therapy; self-compassion; shame; guilt; sexual trauma
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Sexual Trauma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 2 week baseline, CPT + SC (Experimental): Participants in this arm are randomized to a 2-week baseline period with repeated weekly assessment after the initial intake. Following the 2-week baseline, participants are randomly assigned to receive 12 weekly sessions of Cognitive Processing Therapy (CPT), followed by a 3-week return to baseline period, followed by 6 weekly sessions of Self-Compassion Therapy (SC).
  Interventions: Behavioral: Cognitive Processing Therapy; Behavioral: Self-Compassion Therapy
- 2 week baseline, SC + CPT (Experimental): Participants in this arm are randomized to a 2-week baseline period with repeated weekly assessment after the initial intake. Following the 2-week baseline, participants are randomly assigned to receive 6 weekly sessions of Self-Compassion Therapy (SC), followed by a 3-week return to baseline period, followed by 12 weekly sessions of Cognitive Processing Therapy (CPT).
  Interventions: Behavioral: Cognitive Processing Therapy; Behavioral: Self-Compassion Therapy
- 4 week baseline, CPT + SC (Experimental): Participants in this arm are randomized to a 4-week baseline period with repeated weekly assessment after the initial intake. Following the 4-week baseline, participants are randomly assigned to receive 12 weekly sessions of Cognitive Processing Therapy (CPT), followed by a 3-week return to baseline period, followed by 6 weekly sessions of Self-Compassion Therapy (SC).
  Interventions: Behavioral: Cognitive Processing Therapy; Behavioral: Self-Compassion Therapy
- 4 week baseline, SC + CPT (Experimental): Participants in this arm are randomized to a 4-week baseline period with repeated weekly assessment after the initial intake. Following the 4-week baseline, participants are randomly assigned to receive 6 weekly sessions of Self-Compassion Therapy (SC), followed by a 3-week return to baseline period, followed by 12 weekly sessions of Cognitive Processing Therapy (CPT).
  Interventions: Behavioral: Cognitive Processing Therapy; Behavioral: Self-Compassion Therapy

INTERVENTIONS:
Behavioral: Cognitive Processing Therapy — A 12-session cognitive behavioral therapy for posttraumatic stress disorder
Behavioral: Self-Compassion Therapy — A 6-session mindfulness based therapy for posttraumatic stress disorder aimed at enhancing self-compassion

SUMMARY:
Mental contamination-an internal experience of dirtiness evoked in the absence of physical contact with an external source-has been linked to the development and maintenance of posttraumatic stress disorder (PTSD) following exposure to sexual abuse or assault (Adams et al., 2014; Badour et al., 2013; Brake et al., 2017). Mental contamination has been associated with greater PTSD severity (Rachman et al., 2015) and higher elevations in specific PTSD symptom clusters (particularly those of intrusive reexperiencing, negative cognitions/mood, and arousal/reactivity; Brake et al., 2019; Fergus & Bardeen, 2016). Additionally, trauma-related mental contamination has been linked to a number of negative posttraumatic emotions such as shame, guilt, disgust, and anger (Fairbrother & Rachman, 2004; Radomsky & Elliott, 2009) Despite clear and consistent links between mental contamination and problematic posttraumatic outcomes following sexual trauma, there is a dearth of research investigating how existing or promising new interventions for PTSD impact mental contamination.

Cognitive Processing Therapy (CPT) is an efficacious and effective 12-session manualized cognitive-behavioral intervention for PTSD that is considered a gold-standard empirically-supported treatment for PTSD that is recommended by the American Psychological Association (APA, 2017). In addition to PTSD symptom improvement, CPT has also demonstrated benefit for improving feelings of shame and guilt, which are often seen among individuals with trauma-related mental contamination (Nishith et al., 2005; Resick et al., 2002, 2008). Cognitive reappraisal, a primary technique employed in CPT, involves challenging one's view of an emotionally-eliciting situation to alter its emotional impact (Gross & John, 2003). However, some investigators have suggested that cognitive reappraisal may be less effective in targeting moral emotions such as shame, guilt, and self-disgust that are based on an individual's standards and virtues (Finlay, 2015). Self-compassion (SC; i.e., self-directed care and kindness; forgiveness; and feelings of common humanity; Neff, 2003) has been proposed as an alternative method for addressing trauma-related shame and preliminary evidence suggests a 6-session self-compassion intervention may have benefit for reducing both PTSD symptoms and trauma-related shame (Au et al., 2017). Given the centrality of shame, guilt, and self-disgust to the experience of mental contamination, and the fact that mental contamination often arises in response to experiences involving moral violation or betrayal (Millar et al., 2016; Rachman, 2010), a SC intervention for PTSD may also offer promise as a standalone or adjunctive intervention for reducing trauma-related mental contamination. A test of these interventions for their impact on reducing trauma-related mental contamination is needed.

The current study will use Single Case Experimental Design to isolate and evaluate the effects of CPT and SC in reducing both PTSD symptoms and trauma-related mental contamination among individuals with PTSD resulting from sexual trauma.

Aims: 1) explore whether participants demonstrate reductions in mental contamination and PTSD symptoms in response to 12-sessions of CPT or 6-sessions of a SC intervention; 2) evaluate whether presentation of either treatment first yields differences in symptom reduction for PTSD and/or mental contamination symptoms; 3) evaluate whether the addition of the alternative module will enhance reductions in PTSD symptoms and mental contamination; 4) evaluate if such reductions are maintained during follow-up.

Visual inspection analysis and statistical methods will be used to draw conclusions regarding the effects of the interventions on PTSD symptoms and mental contamination.

DETAILED DESCRIPTION:
In this multiple baseline single case experimental design with phase shift, up to 100 participants will be screened to identify 12 eligible individuals to participate in all study procedures. After the baseline assessment, participants will be randomized (1:1 ratio) to either a two or four-week baseline phase (assessment-only). Participants will then be randomized (1:1 ratio) to either a 12-session CPT intervention or a 6-session self-compassion intervention. All participants will complete one orientation session at the beginning of the first treatment phase. Following a second three-week baseline phase, all participants will then shift into the alternate intervention. Participants will be invited to complete a post-treatment and one-month follow-up assessment. In total, participants who take part in this research study will be in this research study for up to 34 weeks and will attend up to 20 in-person study visits.

Individuals interested in participating in this study will complete a phone screening to determine if they are likely to be eligible and can be scheduled for an in-person diagnostic intake to take place at the Stress Trauma and Recovery Research Collaborative (STARRC) within the UK Clinic for Emotional Health (i.e., the PI's research lab space located on Waller Avenue in an office park rented by the University of Kentucky) or via HIPAA compliant Zoom. All participants will be provided with details regarding the phone screen questions and will be required to provide implied consent over the phone before proceeding with the phone screen.

During the intake session, the participant will first be given a written and verbal description of the study and informed consent. The consent form will be presented to the participant on a tablet, or remotely, through REDCap in which they will be asked to provide a digital signature. They may request a paper copy if preferred. If consent is provided, they will be given the option to be emailed a copy. The PI or designated staff will discuss the informed consent form with the participant volunteer. The consent process will take place in a quiet and private room or online via HIPAA compliant Zoom. Participants may take as much time as needed to make a decision about their trial participation and may take the document home if desired. The person obtaining consent will thoroughly explain each element of the document and outline the risks and benefits, alternative treatment(s), and follow-up requirements of the study. Participants will be informed that they can withdraw from the research at any time. Procedures and consent forms will comply with the requirements of the UK Institutional Review Board and Office of Research Integrity's Best Practices for Remote Informed Consent. The experimenter will then complete a consent post-test with participants. If a participant screens out of the study due to a consent capacity issue, any data from that participant that may have been previously collected during the phone screening and/or online surveys will not be used.

Participant privacy will be maintained and questions regarding participation will be answered. No coercion or undue influence will be used in the consent process. No research-related procedures will be performed prior to obtaining informed consent. All signatures and dates will be obtained. A copy of the signed consent will be given to the participant. Signed electronic consents will be maintained and stored through REDCap and will be separated from participant data. We do not have reason to expect that participants are likely to have impaired consent capacity in this study. However, in a previous study our lab conducted where we did have this expectation we included a consent capacity evaluation document and found that we liked using it as an extra check that participants were aware of the study details and what they were agreeing to, and could state back to us in their own words what they could do if they became uncomfortable or decided they wished to take a break, skip sections, or discontinue the study. It is now our lab's standard operating procedure to include this measure in all in-person studies.

Any study personnel member who obtains informed consent from a patient will not serve as that participant's assigned therapist.

Upon referral to the study via the recruitment methods described above, participants will complete a brief telephone screening. The screen will predominantly be conducted by trained undergraduate/post-baccalaureate research/clinic assistants, however the PI, Co-Is, or a supervised graduate students/post-doctoral scholars may also conduct the phone screens. Screening forms for individuals who are deemed to be ineligible for the study will be shredded. Likely eligible participants, determined by the phone screen, will be invited to attend the intake in-person in the PI's research lab at the Clinic for Emotional Health or via HIPAA-compliant video conferencing service (i.e., Zoom via the UK HealthCare portal). As described above (see "Informed Consent" section), a study assessor (i.e., doctoral students in clinical psychology/post-doctoral scholar/PI/Co-Is) will review study procedures with potential participants and ask them to provide their informed consent. After informed consent is provided, an interview-based diagnostic assessment will be administered in order to confirm clinical inclusion/exclusion criteria. This assessment visit will be video or audio-recorded provided participants give their consent for this.

Next, participants will be asked to complete a battery of self-report questionnaires, which will assess symptoms of anxiety/depression, level of functioning (e.g., quality of life), experiential avoidance, self-compassion, and perceptions of how their history of sexual trauma have impacted their life. Those who are deemed ineligible after this assessment will be withdrawn.

Eligible participants will then be randomized to either a two- or four-week baseline where they will complete weekly measures of PTSD symptoms mental contamination, trauma-related shame and guilt, and symptoms of anxiety/depression. This battery will be repeated each week during therapy sessions, along with additional post-session ratings about treatment credibility and therapeutic alliance. Participants will then be randomly assigned to one of two treatment orders (CPT, SC or SC, CPT) and will be scheduled for their next study session either in-person or via HIPAA compliant Zoom. All participants will first be scheduled for a therapy orientation session prior to beginning either CPT or SC. The therapy orientation session will be used to develop rapport between the therapist and participant, and will involve an interview to assess for details of the index traumatic event and experiences of trauma-related mental contamination. Following completion of each treatment (12 or 6 sessions), participants will be asked to provide satisfaction ratings and written qualitative feedback on their experience with the treatment they received. Participants will then enter a second three-week return to assessment period where they will continue to complete questionnaires weekly before beginning the second treatment module. Participants will also complete a post-treatment questionnaire packet and continue to track their symptoms weekly for three weeks following the conclusion of treatment via self-report.

All therapy sessions will last for approximately 60-90 minutes in duration. It is important to note that the therapeutic strategies involved in both treatments are all common, evidence-based cognitive-behavioral- or mindfulness-based strategies. The treatments involve reading from an established manual (Cognitive Processing Therapy for PTSD or Compassion-Based Therapy for Trauma-Related Shame and Posttraumatic Stress) and completing homework assignments outside of the treatment session. These treatment sessions will be audio- or video-recorded provided participants give their consent for this; this will allow study staff to rate sessions for fidelity to the protocol and will be used for clinical supervision.

All self-report questionnaires will be completed online via REDCap. This survey platform is designed specifically for collection of research data, and therefore meets the privacy standards imposed on health care records by the Health Insurance Portability and Accountability Act (HIPAA). Questionnaires will be completed on-site using a study iPad or participants will be sent a link via email to complete the survey batteries during their own time. Finally, although we anticipate that most patients will prefer to complete these measure electronically, we can provide paper and pencil versions of the questionnaires if requested.

Data collection will be accomplished via phone screening questions, diagnostic interview, and self-report questionnaires attached below. Through these measures we will collect data regarding participants' experiences with psychological symptoms, life functioning, and treatment satisfaction.

The measures will be administered according to the following schedule:

Intake and Final Treatment Sessions:

Diagnostic Interview for Anxiety, Mood, and Obsessive-Compulsive and Related Neuropsychiatric Disorders (DIAMOND) interview (Only at Intake) Columbia-Suicide Severity Rating Scale (CSSRS) with SAFE-T Risk Assessment Demographics (Only at Intake) PTSD Checklist for DSM-5 (PCL-5) - Weekly Posttraumatic Experience of Mental Contamination (PEMC) - Weekly Trauma-Related Symptom Inventory (TRSI) - Weekly Trauma-Related Guilt Inventory (TRGI) - Weekly Overall Depression Severity and Impairment Scale (ODSIS) - Weekly Overall Anxiety Severity and Impairment Scale (OASIS) - Weekly Centrality of Events Scale (CES) Self-Compassion Scale (SCS) Obsessive Compulsive Inventory-Revised (OCI-R) Brief Experiential Avoidance Questionnaire (BEAQ) Quality of Life Enjoyment and Satisfaction Questionnaire-Short Form (Q-LES-Q) Patient Satisfaction Form (final treatment sessions only)

Treatment Orientation Session:

Treatment Services Tracking Form (Intake only) Trauma Interview

Pre-Session (Weekly):

PCL-5 - Weekly PEMC - Weekly TRSI - Weekly TRGI - Weekly CSSRS - Weekly (in-person sessions only) Treatment Services Tracking Form - Weekly (in-person sessions only)

Post-Session (Weekly):

ODSIS - Weekly OASIS - Weekly Helping Alliance Questionnaire-II (HAQ-II) - Patient and Therapist CEQ (post-1st treatment sessions only)

The goal of Aim 1 is to collect descriptive information regarding prevalence of trauma history and PTSD, perceptions of connections between trauma history and substance use, and interest in trauma-informed treatment. This information will be utilized to a) support the feasibility of a future grant application and b) identify potential patients for the treatment portion of the study.

Though the primary focus of Aim 2 is to collect data regarding feasibility, acceptability, and patient feedback regarding areas of modification to inform a future grant proposal, we plan to utilize a randomized, nonconcurrent multiple baseline design across participants (Barlow et al., 2009; Kazdin, 2011). This is a form of single-case experimental design that provides a time and cost-effective method of evaluating initial efficacy or effectiveness of an intervention while controlling for the passage of time and repeated assessment in small numbers of patients. Patients will be randomized to either a 2- (n=3) or 4-week (n =3) baseline assessment phase where weekly self-report measures will be completed prior to initiating each treatment. Randomizing to varying baseline periods enables assessments of whether symptoms change (only or more rapidly) when the intervention is applied (i.e., each participant acts as their own control). Participants will also be randomly assigned to the order that they receive the treatment, with a 3-week return to baseline between treatments to allow us to examine how symptoms change within each intervention period. This design allows for causal inferences and controls for many threats to internal validity. Consistent with established guidelines, quantitative data analysis will primarily be conducted via visual inspection of graphed data within- and between-subjects to evaluate the magnitude and rate of change across the baseline and treatment phases (Barlow et al., 2009; Kazdin, 2011). This will be supplemented by examining within-person mean difference effect sizes for each outcome using a d-statistic developed for single case designs and calculating the percentage of patients who evidence reliable change on symptom measures (Jacobson & Truax, 1991; Shadish et al., 2014).

ELIGIBILITY:
Inclusion Criteria:

* individuals with a history of sexual trauma meeting past-month diagnostic criteria for PTSD (meeting diagnostic status on the DIAMOND and score greater than or equal to 36 on the PCL-5) and
* reporting current experiences of trauma-related mental contamination (greater than or equal to 10 on the PEMC).
* 18 years of age or older
* fluent in English
* Patients on psychotropic medications will be included if they have been maintained on a stable dose for at least 4 weeks prior to beginning the study and are willing to maintain a stable dosage throughout the study period; this procedure allows for a broader range of participants and avoids having outcomes assessment confounded by the initiation of medication during treatment.
* Finally, patients must be willing to refrain from additional trauma-related treatment for the duration of the study.

Exclusion Criteria:

* We will exclude individuals diagnosed with psychological conditions that may be better addressed by alternative treatments; these conditions include
* psychotic disorders
* dissociative identity disorder
* unmanaged (i.e., unmedicated or currently experiencing a manic/hypomanic episode) bipolar disorder
* bulimia nervosa
* anorexia nervosa
* imminent risk of suicide (i.e., intent/plan)
* severe substance use disorders.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2020-09-10 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
PTSD Checklist for DSM-5 (PCL-5) | Change in prior week symptom severity assessed from 3 or 5 weeks prior to beginning treatment (intake + baseline), compared to weekly during treatment, compared to 3 weeks between treatments, and compared to 3 weeks after completing the second treatment
  Change in Posttraumatic Stress Disorder Symptom Severity
Posttraumatic Experience of Mental Contamination (PEMC) | Change in prior week symptom severity assessed from 3 or 5 weeks prior to beginning treatment (intake + baseline), compared to weekly during treatment, compared to 3 weeks between treatments, and compared to 3 weeks after completing the second treatment
  Change in Severity of Mental Contamination Symptoms

SECONDARY OUTCOMES:
Trauma-Related Shame Inventory (TRSI) | Change in prior week symptom severity assessed from 3 or 5 weeks prior to beginning treatment (intake + baseline), compared to weekly during treatment, compared to 3 weeks between treatments, and compared to 3 weeks after completing the second treatment
  Change in Severity of Trauma-Related Shame
Trauma-Related Guilt Inventory (TRGI) | Change in prior week symptom severity assessed from 3 or 5 weeks prior to beginning treatment (intake + baseline), compared to weekly during treatment, compared to 3 weeks between treatments, and compared to 3 weeks after completing the second treatment
  Change in severity of Trauma-Related Guilt

CONTACTS AND LOCATIONS:
Overall Officials: Christal L Badour, PhD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky Clinic for Emotional Health (CEH), Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication and are de-identified will be shared with investigators upon request.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Data will be shared upon request from investigators beginning immediately after publication
Access Criteria: Researchers who provide a methodologically sound proposal.